CLINICAL TRIAL: NCT04484415
Title: A Double Blind, Prospective, Randomized, Placebo Controlled, Multi-center Phase 3 Study to Evaluate Efficacy and Safety of Cevira® in Patients With Cervical Histologic High-grade Squamous Intraepithelial Lesions (HSIL)
Brief Title: Efficacy and Safety of Cevira® in Patients With Cervical Histologic High-grade Squamous Intraepithelial Lesions (HSIL)
Acronym: APRICITY
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Asieris MediTech (Hong Kong) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Jiangsu Yahong Meditech Co., Ltd aka Asieris (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YHGT-CEV-R1
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Cervical Intraepithelial Neoplasia Grade 2/3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cevira® treatment (Experimental): The Cevira® treatment is an integrated combination of drug and device
  Interventions: Combination Product: Cevira®
- Placebo ointment (Placebo Comparator): The placebo ointment contains only vehicle, and is similar in appearance and consistence as the Cevira® ointment. The placebo device is identical in appearance as the Cevira® device, but does not provide light.
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Combination Product: Cevira® — The device is a single-use, disposable, LED-based red light source. The device will automatically switch on the light 5 hours after administration, and provide continuous photoactivation of 125 J/cm2 over 4.6 hours before automatically shutting down.
  Arms: Cevira® treatment
Combination Product: Placebo — The placebo device is identical in appearance as the Cevira® device, but does not provide light.
  Arms: Placebo ointment

SUMMARY:
A double blind, prospective, randomized, placebo controlled, multi-center phase 3 study to evaluate efficacy and safety of Cevira® in patients with cervical histologic high-grade squamous intraepithelial lesions (HSIL).

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of Cevira® compared to placebo in treatment of patients with cervical histologic HSIL.A total of 384 subjects will be enrolled globally, among which, 300 subjects of them will be enrolled in China.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-confirmed HSIL histology determined by a panel of 3 pathologists from a central laboratory in each region (China, US, and Europe);
2. Adequate colposcopy including:

   1. visualization of entire cervical transformation zone including the squamocolumnar junction
   2. visualization of entire lesion margin
3. Colposcopically visible lesion after biopsy, before treatment (Note: To ensure a colposcopically visible lesion after biopsy, the lesion should cover approximately 15% of the uterine cervix before biopsy)
4. Average sized uterine cervix suitable for application of the Cevira® device
5. Use of adequate birth control until completion of the 6 month assessment visit
6. Age 18 or older (Note: Patients aged 18-20 should not be actively recruited)
7. Signed written informed consent

Exclusion Criteria:

1. Biopsy-confirmed HSIL (CIN3) histology with a total lesion area covering more than half of the uterine cervix area
2. Invasive cervical cancer
3. Adenocarcinoma in situ, or other glandular intraepithelial lesions
4. Lesion(s) extending to the cervical canal (as clinically indicated and whether to perform endocervical curettage [ECC] test at the discretion of the investigators)
5. Lesion(s) extending to the vaginal vault
6. Current severe pelvic inflammatory disease, severe cervicitis, or other severe gynecological infection as per colposcopy and clinical examination
7. Vaginal bleeding at time of treatment at the discretion of the investigator
8. Pregnancy
9. Nursing
10. Childbirth or miscarriage within six weeks of enrolment
11. Patients who previously received surgical treatment, have incomplete cervical structure and have recurrent HSIL; or patients who received other treatment after the confirmed diagnosis of HSIL
12. History of toxic shock syndrome
13. Known or suspected porphyria
14. Known allergy to hexaminolevulinate or similar compounds (e.g. methyl aminolevulinate or aminolevulinic acid)
15. Known allergy to silicone
16. Use of heart pacemaker
17. Participation in other therapeutic clinical trials using investigational agents either concurrently or within the last 30 days
18. Patients that in the investigator's opinion are not suitable for participation
19. Patient is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the study

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of responders at 6 months after first treatment | 6 months
  A responder is defined as follows:
  * Normal histology; or
  * LSIL histology and clearance of baseline HPV

SECONDARY OUTCOMES:
The proportion of HPV positive patients with clearance of baseline HPV at 6 months after first treatment. | 6 months
  The proportion of HPV positive patients with clearance of baseline HPV at 6 months after first treatment.
The proportion of HPV16 positive patients with clearance of HPV16 at 6 months after first treatment. | 6 months
  The proportion of HPV16 positive patients with clearance of HPV16 at 6 months after first treatment.
The proportion of HPV16 and/or HPV18 positive patients with clearance of baseline HPV at 6 months after first treatment. | 6 months
  The proportion of HPV16 and/or HPV18 positive patients with clearance of baseline HPV at 6 months after first treatment.
The proportion of patients with histologic regression, defined as LSIL or normal histology, at 6 months after first treatment. | 6 months
  The proportion of patients with histologic regression, defined as LSIL or normal histology, at 6 months after first treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jinghe Lang, MD,PhD, Principal Investigator — Peking Union Medical College Hospital; John Zhuang, PhD, Study Chair — Asieris MediTech (Hong Kong) Co., Ltd.
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen F, Novak Z, Dannecker C, Mokras C, Sui L, Zhang Y, You Z, Han L, Lang J, Hillemanns P. Multicentre, prospective, randomised controlled trial to evaluate hexaminolevulinate photodynamic therapy (Cevira) as a novel treatment in patients with high-grade squamous intraepithelial lesion: APRICITY phase 3 study protocol. BMJ Open. 2022 Jun 6;12(6):e061740. doi: 10.1136/bmjopen-2022-061740. PMID 35667715